CLINICAL TRIAL: NCT06047717
Title: The Impact of Vision Loss on Naturalistic Behavior and Navigation in Virtual Reality
Brief Title: Vision Loss Impact on Navigation in Virtual Reality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Rochester Institute of Technology (Other)
Responsible Party: Principal Investigator, Krystel Huxlin, James V. Aquavella Professor of Ophthalmology, Associate Chair for Research, Dept. Ophthalmology, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00008669
Record Dates: First submitted 2023-09-08; First posted 2023-09-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Stroke, Ischemic; Quadrantanopia; Hemianopsia, Homonymous; Hemianopia, Homonymous; Hemianopia; Hemianopsia; Occipital Lobe Infarct; Visual Field Defect, Peripheral; Vision Loss Partial; Quadrantanopsia; Stroke Hemorrhagic
Keywords: Occipital stroke; Vision loss after stroke; Vision recovery; Vision restoration; Partial vision loss; Homonymous quadrantanopsia; Homonymous quadrantanopia; stroke
MeSH Terms: conditions — Ischemic Stroke; Hemianopsia; Hemorrhagic Stroke; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) Driving Task: Cortically Blind Cohort (Experimental): Persons who have sustained cortical blindness will perform a driving task in VR, in which they must steer through a series of parameterized turns while maintaining their virtual vehicle centered between the two red lines delineating the "road" edge.
  Interventions: Other: Virtual Reality Driving Task
- Virtual Reality (VR) Driving Task: Healthy Control Cohort (Experimental): Healthy controls with no vision loss will perform a driving task in VR, in which they must steer through a series of parameterized turns while maintaining their virtual vehicle centered between the two red lines delineating the "road" edge.
  Interventions: Other: Virtual Reality Driving Task

INTERVENTIONS:
Other: Virtual Reality Driving Task — Participants will steer a virtual car with the goal of staying in the center of a single-lane roadway while traveling at a constant speed of 26.6 m/s (approximately 60 miles/hr). The roadway alternates between a series of straights and turns of different radii to both the left and the right. This allows for careful control of task difficulty, and for the repeated presentation of specific conditions across multiple "trials" (i.e. turns in the road) in a randomized order. In addition, the density of the visual texture elements in the virtual environment that provide optic flow (OF) signal is also varied. The low-density OF condition has no road texture or foliage, and only the solid road edges on a flat-black ground plane. The medium-density OF condition has sparse textural elements distributed on the ground plane, and the high-density OF condition has high density road texture and a canopy of road-side trees that provide texture extending far above the horizon.

SUMMARY:
The purpose of this research is to better understand the impact of cortically-induced blindness (CB) and the compensatory strategies subjects with this condition may develop on naturalistic behaviors, specifically, driving. Using a novel Virtual Reality (VR) program, the researchers will gather data on steering behavior in a variety of simulated naturalistic environments. Through the combined use of computer vision, deep learning, and gaze-contingent manipulations of the visual field, this work will test the central hypothesis that changes to visually guided steering behaviors in CB are a consequence of changes to the visual sampling and processing of task-related motion information (i.e., optic flow).

ELIGIBILITY:
Cortically Blind Group:

Inclusion Criteria:

* Residents of the United States or Canada
* Presence of one-sided stroke or stroke-like damage to primary visual cortex or its immediate afferent white matter sustained within the specified age range of 21 - 75 years (verified by MRI and/or CT scans)
* Reliable visual field defects in both eyes (homonymous defects) as measured by Humphrey or equivalent perimetry.
* Willing, able, and competent to provide their own informed consent
* Cognitively able, responsible to understand written and oral instructions in English
* Emmetropic or else wear corrective contact lenses inside the virtual reality headset

Exclusion Criteria:

* Those who have never driven or earned a drivers' license
* Past or present ocular disease interfering with visual acuity
* Best corrected visual acuity (BCVA) worse than 20/40 in either eye
* Sustained damage to the dorsal lateral geniculate nucleus
* Presence of diffuse, whole-brain degenerative processes
* Presence of brain damage deemed by study staff to potentially interfere with outcome measures
* History of traumatic brain injury
* Documented history of drug/alcohol abuse
* Diagnosis of cognitive or seizure disorders
* Diagnosis of one-sided attentional neglect

Control Group:

Inclusion Criteria:

* Normal or corrected-to-normal vision, who are between the ages of 21 and 75 years of age, roughly matched to the age of CB subjects enrolled above
* Competent and responsible, as determined by the Principal Investigator
* Willing, able, and competent to provide their own informed consent
* Normal cognitive abilities, be able to understand written and oral instructions in English
* Emmetropic or else wear corrective contact lenses inside the virtual reality headset

Exclusion Criteria:

* Subjects who have never driven or earned a drivers' license
* BCVA worse than 20/40 in either eye
* Presence of vision loss from ocular diseases or disorders
* Presence of a visual field defect
* Inability to wear corrective contact lenses inside the virtual reality helmet if required to see clearly
* Subjects with a history of neurological disorders
* Subjects with a history of TBI
* Persons who lack the competence or are otherwise unable to perform the visual testing as directed.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Virtual Reality (VR) Lane Deviation / Offset | Day 0
  Virtual lane offset is a measure of driving accuracy, which involves computing the divergence (in virtual meters) from the center of the single-lane virtual roadway, relative to the position of the driver's head and averaged over the duration of each turn. The researchers will compare the variance of lane offset in virtual meters between Cortically Blind (CB) and control subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States